CLINICAL TRIAL: NCT06411210
Title: Obesity Complicating Type 1 Diabetes in Young Adults: Physiology and Impact of GLP-1 Analogue Anti-obesity Treatment on Cardiometabolic Risk Factors
Brief Title: Obesity Complicating Type 1 Diabetes: GLP-1 Analogue Anti-obesity Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Michelle Van Name, Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000035452; 1R01DK134398-01A1 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Diabetes type1; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Participants in this arm will receive semaglutide (escalated to 2.4mg or max tolerated dose) weekly for 12 months. Then a 4 week wean period plus 2 weeks as needed insulin titration.
  Interventions: Drug: Semaglutide Pen Injector
- Placebo (Placebo Comparator): Participants in this arm will receive a matched placebo weekly for 12 months. Then a 4 week wean period plus 2 weeks as needed insulin titration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Pen Injector — Escalated to 2.4mg or max tolerated dose
  Arms: Semaglutide
Drug: Placebo — Matched placebo.
  Arms: Placebo

SUMMARY:
More than 40% of young adults with type 1 diabetes (T1D) also have overweight or obesity. Each of these diagnoses increase the risk of adverse cardiovascular events. GLP-1 analogues are anti-obesity medications that are cardioprotective in adults with type 2 diabetes, however evaluation of these agents in people with T1D has been limited to glycemic outcomes. Investigators aim to study the impact of GLP-1 analogue obesity treatment on markers of cardiometabolic risk in young adults with T1D and obesity.

DETAILED DESCRIPTION:
This proposal will address critical knowledge gaps of understanding potential salutary effects of GLP-1 analogue anti-obesity treatment with weekly semaglutide 2.4 mg on cardiometabolic risk factors in young adults with T1D and obesity, the group of people with T1D at greatest risk for future cardiovascular disease. Investigators aim to examine the impact of 12 months of treatment with weekly semaglutide 2.4 mg compared to placebo on abdominal adipose tissue distribution, glucose metabolism and postprandial atherosclerotic lipoproteins in young people with T1D and obesity.

This is a single-center, parallel group, double-blinded, placebo controlled, randomized clinical trial. After informed consent procedures, participants will complete four assessments: 1) Abdominal MRI to evaluate abdominal adipose partitioning, 2) Euglycemic hyperinsulinemic clamp with isotope tracer enhancement to evaluate gluconeogenesis and glucose, glycerol, and b-hydroxybutyrate turnover to assess measures of insulin resistance, 3) DEXA scan to evaluate total body composition, and 4) a High-fat mixed meal tolerance test to evaluate postprandial lipemia. After completing these baseline measures, participants will be randomized in a 2:1 ratio to receive weekly injected semaglutide (escalated to 2.4 mg or maximum tolerated dose) or placebo to treat obesity for 52 weeks. At 52 weeks, participants will repeat the baseline tests. They will then complete a wean off of study drug (up to 4 weeks) and 2 weeks of additional monitoring for insulin titration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years with T1D whose BMI meets FDA approval criteria for anti-obesity pharmacotherapy (BMI ≥30 kg/m2 alone or BMI ≥27 kg/m2 with a weight-related comorbidity)
* Clinical diagnosis of T1D
* Diabetes duration diagnosed ≥ 12 months ago
* HbA1c ≤10% at screening and within the past 90 days
* Stable reported insulin dosing in the past 90 days (within 15%)
* Stable reported BMI in the past 90 days (within 5%)
* Ability to provide written informed consent before any trial-related activities
* Use of real-time continuous glucose monitoring and planned continued use
* Females and males of childbearing potential willing to use highly effective methods of contraception for at least 1 month prior to randomization and agreement to use such a method during study participation and for 2 months after the last dose of study medication administration: Combined estrogen-progestogen contraception including: oral, intravaginal, transdermal (patch), Progestogen-only contraception: oral, injectable or implantable, Placement of an intrauterine device or intrauterine system, Bilateral tubal occlusion (fallopian tubes are blocked), Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate), or Complete sexual abstinence from male-female sex)
* Stated willingness to comply with all study procedures, medication regimen, and availability for the duration of the study
* Participants cannot be randomized if any laboratory safety parameter at screening is outside the below extended laboratory ranges. For randomization, participants should have

  1. Creatinine <1.0mg
  2. Triglycerides (<400 mg/dl)
  3. ALT <3.5 times the upper normal limit (UNL)

Exclusion Criteria:

* Use of adjunctive diabetes therapies or anti-obesity medications (including any GLP-1 agonist) currently or within the past 6 months.
* Insulin dosing <0.5 units/kg/day
* Current psychiatric conditions impacting weight, including known eating disorders
* Contraindications to study medications, including:

  * Personal history of pancreatitis, renal impairment, or known liver disease other than non-alcoholic hepatic steatosis
  * Personal or family history of medullary thyroid cancer or Multiple Endocrine Neoplasia Type 2
  * Known or suspected allergy to semaglutide, excipients, or related products.
* Use of lipid lowering medications other than statins and omega-3 products
* Previous randomization in this trial. Participants who enrolled but did not randomize can be re-screened. Potential reasons for enrolment without randomization include scheduling conflicts for the baseline studies, or for females, not yet meeting the highly effective methods of contraception criteria.
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures
* Diabetic ketoacidosis in the past 6 months
* Not meeting MRI safety criteria or claustrophobia preventing participation in the MRI
* Anemia or known hematologic condition impacting HbA1c reading, or another medical condition that precludes participation.
* Treatment with another investigational drug or other intervention within the past 1 month
* Subjects with a PHQ-9 score >15 or those found to have a lifetime history of suicide attempts, or suicidal ideation within the past 3 months on the C-SSRS
* Corn allergy
* Subjects with severe hypoglycemia requiring hospitalization in the past 3 months
* Clinically significant gastroparesis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in VAT/(VAT+SAT) from baseline to 12 months | baseline and 12 months
  Measured as VAT/Subcutaneous Adipose Tissue + VAT changes over 1 year.
Change in hepatic insulin resistance from baseline to 12 months | baseline and 12 months
  Hepatic insulin resistance, measured by serum concentration of beta-hydroxybutyrate (surrogate marker of acetyl-CoA, which regulates gluconeogenesis), changes over 1 year.
Change in triglycerides from baseline to 12 months | baseline and 12 months
  Change in triglycerides after a high-fat mixed meal tolerance test, expressed as the total Area Under the Curve (AUCTG) over 6 hours from baseline to 1 year.

SECONDARY OUTCOMES:
Change in weight from baseline to 12 months | baseline and 12 months
  Mean change in weight (kilograms) assessed using a scale
Change in percent body fat from baseline to 12 months | baseline and 12 months
  Mean change in percent body fat assessed using DEXA scan measurements
Change in BMI from baseline to 12 months | baseline and 12 months
  Mean change in BMI calculated using measured height and weight.
Change in mean glucose concentration | baseline and 12 months
  Change in mean glucose concentration. Data collected as available using participant's personal clinical continuous glucose monitor.
Mean time in normal glucose range | baseline and 12 months
  Mean time in normal glucose range. Range=70-180 mg/dl and 3.9-10 mmol/L. Data collected as available using participant's personal clinical continuous glucose monitor.
Mean time in level 1 and 2 hyperglycemia, high range | baseline and 12 months
  Mean time in level 1 and 2 hyperglycemia. Range= >180, >250 mg/dL and >10, >13.9 mmol/L. Data collected as available using participant's personal clinical continuous glucose monitor.
Mean time in level 1 and 2 hyperglycemia, low range | baseline and 12 months
  Mean time in level 1 and 2 hyperglycemia. Range= <70, <54 mg/dL and <3.9, <3.0 mmol/L. Data collected as available using participant's personal clinical continuous glucose monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Van Name, MD, Principal Investigator — Yale University
Locations (1):
- Yale Pediatric Diabetes Center, Adult and Children's Progam, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No